CLINICAL TRIAL: NCT06259188
Title: Investigation of the Effectiveness of Personalized Breathing Exercise Device in Patients With COPD
Brief Title: Effectiveness of Personalized Breathing Exercise Device in Patients With COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Biruni University (Other); The Scientific and Technological Research Council of Turkey (Other); Istanbul University (Other)
Responsible Party: Principal Investigator, Ozge Ertan, Physiotherapist MSc, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1001
Record Dates: First submitted 2024-01-19; First posted 2024-02-14 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; Inspiratory Muscle Training; Expiratory Muscle Training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Breathing Exercise Device Group (Experimental): In the personalized respiratory exercise device group, the initial pressure load will be set to the resistance level corresponding to 40% of the MIP and MEP measurements. Participants will be asked to rest following 5 breathing cycles and repeat the training for 10 sets. In each set, there will be a one-minute rest break between repetitions. Participants will be able to practice both inspiratory and expiratory respiratory muscle training in a single breathing cycle. As the progression progresses, the perceived exertion level will be increased by 5-10% on a weekly basis, to be in the range of 4-6 according to the Modified Borg scale.
  Interventions: Device: Personalized Breathing Exercise Device
- Respiratory Muscle Training Group (Active Comparator): Respiratory muscle training will be done with Threshold® IMT and Threshold™ PEP devices. Training intensity will be set to 40% of MIP and MEP measurements in the first week. For inspiratory muscle training, participants will be asked to rest after 5 breathing repetitions and repeat the training for 10 sets. Participants will be asked to rest after 5 exhalation repetitions for expiratory muscle training and repeat the training for 10 sets. In each set, there will be a one-minute rest break between repetitions. As the progression progresses, the perceived exertion level will be increased by 5-10% on a weekly basis, to be in the range of 4-6 according to the Modified Borg scale. At this point, if the training threshold exceeds the upper pressure limits of Threshold® IMT + Threshold™ PEP devices, the training intensity will continue at the upper limit.
  Interventions: Device: Respiratory Muscle Training Device

INTERVENTIONS:
Device: Respiratory Muscle Training Device — In the both groups the initial pressure load will be set to the resistance level corresponding to the 40% of the MIP and MEP measurement. Participants will be asked to rest following 5 breathing cycles and repeat the training for 10 sets. In each set, there will be a one-minute rest break between repetitions. In breathing exercise device group participants will be able to practice both inspiratory and expiratory respiratory muscle training in a single breathing cycle. In IMT+EMT group, patients will be able to practice different to device. As the progression progresses, the perceived exertion level will be increased by 5-10% every week, to be in the range of 4-6 according to the Modified Borg scale.
  Arms: Respiratory Muscle Training Group
Device: Personalized Breathing Exercise Device — Personalized Breathing Exercise Device
  Arms: Personalized Breathing Exercise Device Group

SUMMARY:
The current "Global Initiative for Chronic Obstructive Lung Diseases" (GOLD) guideline emphasizes that pulmonary rehabilitation should be recommended to all chronic obstructive pulmonary disease (COPD) patients from Stage II onwards. Respiratory muscle training applied to individuals with COPD is an important part of pulmonary rehabilitation due to its benefits such as improving pulmonary function and respiratory muscle strength, reducing the severity of dyspnea, and increasing exercise capacity and quality of life. Although there is sufficient evidence in the literature about the benefits of IMT in individuals with COPD. There is little evidence showing the effects of EMT. Studies show that isolated IMT and EMT are effective in increasing respiratory muscle strength, endurance and exercise capacity. Results from a limited number of studies show that combined training of IMT and EMT is superior compared to isolated IMT or isolated EMT in improving exercise capacity and dyspnea. Incentive spirometers, with their different mechanical properties, are low-cost respiratory exercise devices that are widely used in the early postoperative period, lung diseases, long-term bed rest and in situations where it is necessary to maintain or increase the ventilation ability of the lung, but they do not apply any resistance to the respiratory muscles. In the pulmonary rehabilitation guidelines published by the American Thoracic Society (ATS) and the European Respiratory Society (ERS), the necessity of using devices that apply resistance to the respiratory muscles to strengthen the respiratory muscles is underlined. The personalized respiratory exercise device will be a device that has the clinical features of an incentive spirometer and respiratory muscle training devices (inspiratory and expiratory) and can be personalized according to the desired purpose. With the same device, patients will be able to both improve lung ventilation, such as an incentive spirometer, and strengthen their respiratory muscles.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD by a pulmonologist according to GOLD 2022 diagnostic criteria (GOLD, 2022) and in classes B, C and D according to GOLD
* Followed for at least 6 months
* Clinically stable patients without exacerbations or infections

Exclusion Criteria:

* Patients with a history of spontaneous or trauma-related pneumothorax
* Patients with middle ear-related pathologies (such as tympanic membrane rupture, otitis)
* Orthopedic and neurological problems that may interfere with exercise training
* Changes in medical treatment during the study
* Patients with unstable concomitant cardiac disease
* Patients who have been involved in another pulmonary rehabilitation program within the last 6 months
* Insufficient cooperation

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-05-29 (Estimated); Study Completion 2025-05-29 (Estimated)

PRIMARY OUTCOMES:
Maximal static inspiratory mouth pressure | 1 week-8 week
  Measurement will be made with a respiratory muscle strength measuring device. MIP: maximal inspiratory pressure
Maximal static expiratory mouth pressure | 1 week-8 week
  Measurement will be made with a respiratory muscle strength measuring device. MEP: maximal expiratory pressure

SECONDARY OUTCOMES:
Respiratory Functions FEV1 | 1 week-8 week
  Pulmonary function test: FEV1 L and %
Respiratory Functions FVC | 1 week-8 week
  Pulmonary function test: FVC L and %
Respiratory Functions FEV1/FVC | 1 week-8 week
  Pulmonary function test: FEV1/FVC%
Respiratory Functions PEF | 1 week-8 week
  Pulmonary function test: PEF L/S and %
Diffusion Capacity | 1 week-8 week
  Pulmonary function test: DLCO%
Exercise capacity | 1 week-8 week
  Spiropalm six minute walk test
Activities of daily living | 1 week-8 week
  London Chest Activities of Daily Living Scale (LCADL): Perceived dyspnea while performing activities of daily living is scored between 0-5. A high score indicates greater disability in performing ADLs. The minimum total score 0 and maximum total score is 75.
Activity Status | 1 week-8 week
  Duke Activity Status Index: The Duke Activity Status Index (DASI) is a patient-reported estimate of functional capacity, maximal oxygen consumption (VO2 max) and maximum metabolic equivalent of tasks (METs). The DASI questionnaire produces a score between 0 and 58.2 points
Device ease of use | 8 week
  5-Likert Scale: Scoring will be determined as 1- "very difficult to use" and 5- "very easy to use".

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Ertan, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)